CLINICAL TRIAL: NCT06567782
Title: A Phase 2, Open Label, Randomized Study of Neoadjuvant Dostarlimab Plus CAPEOX Versus CAPEOX in Participants With Previously Untreated T4N0 or Stage III MMRp/ MSS Colon Cancer
Brief Title: A Study of Neoadjuvant Dostarlimab Plus Capecitabine Plus Oxaliplatin (CAPEOX) Vs CAPEOX With Previously Untreated T4N0 or Stage III Mismatch Repair Proficient (MMRp)/Microsatellite Stable (MSS) Colon Cancer
Acronym: AZUR-4
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222892; 2024-513441-36 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms, Colon
Keywords: Colon cancer; MMRp; MSS; Dostarlimab; CAPEOX; Neoadjuvant; GSK4057190A; TSR-042; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dostarlimab plus CAPEOX (Experimental): Participants will receive dostarlimab plus CAPEOX (chemotherapy).
  Interventions: Biological: Dostarlimab; Drug: CAPEOX
- CAPEOX (Active Comparator): Participants will receive CAPEOX (chemotherapy).
  Interventions: Drug: CAPEOX

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
  Other Names: GSK4057190A; TSR-042
  Arms: Dostarlimab plus CAPEOX
Drug: CAPEOX — CAPEOX chemotherapy consisting of capecitabine and oxaliplatin will be administered.

SUMMARY:
The main goal of this study is to test a new treatment approach for colon cancer. The treatment involves dostarlimab along with a specific type of chemotherapy called CAPEOX (short for "capecitabine + oxaliplatin") to check if using these two together works better than using just CAPEOX by itself. This treatment is given before any surgery takes place; a method referred to as "neoadjuvant therapy." . The aim is to see if this new approach can show early signs of effectiveness in treating participants with a specific type of colon cancer known as mismatch repair proficient/ microsatellite stable (MMRp/MSS), where the cells have normal repair systems and stable DNA sequences. This study will also look at specific signs in the blood and tumor to see if they can help predict how well the treatment is working. This could help better understand how dostarlimab contributes to the response of the disease to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has untreated pathologically confirmed colon adenocarcinoma
* Has resectable colon adenocarcinoma defined as clinically T4N0 or Stage III
* Has a tumor demonstrating the presence of either-

  1. MMR status: MMR status must be assessed by Immunohistochemistry (IHC) for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where all proteins are present indicates MMRp; MMR status may be determined local laboratory; or
  2. MSS or Microsatellite Instability-L (MSI-L) phenotype as determined by polymerase chain reaction (PCR) or by tissue next generation sequencing (NGS), determined by local laboratory
* Provides fresh tumor tissue obtained during either the pre-screening or screening period via colonoscopy performed per procedure manual. Tissue biopsy is required
* Is willing to use adequate contraception male and/or female participants
* Has an Eastern Cooperative Oncology Group - Performance status (ECOG-PS) of 0 or 1
* Has adequate organ function

Exclusion Criteria:

* Has distant metastatic disease
* Has received prior medical therapy (chemotherapy, immunotherapy, biologic, or targeted therapy), radiation therapy or surgery for management of colon cancer
* Has, in the investigator's opinion, a tumor that is not amenable to surgery or has any other contraindication to surgery
* Has experienced any of the following with prior immunotherapy: any imAE ≥ Grade 3, immune-mediated severe neurologic events of any-grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade [Stevens-Johnson Syndrome (SJS), Toxic Epidermal Necrolysis (TEN), or Drug rash with eosinophilia and systemic symptoms (DRESS) syndrome], or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary
* Has any history of interstitial lung disease or immune-related pneumonitis
* Has a history or current evidence of any medical condition, therapy, or laboratory abnormality that might confound the study results, interfere with their participation for the full duration of the study intervention, or indicate it is not in the best interest of the participant to participate, in the opinion of the investigator
* Is considered, in investigator's opinion, a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active infection requiring systemic therapy
* Has received treatment with an investigational agent within [4 weeks] of the first dose of study intervention
* Is pregnant or breastfeeding
* Has a history of severe allergic and/or anaphylactic reactions to chimeric, human, or humanized antibodies, fusion proteins, or known allergies to dostarlimab, or its excipients, or any components of CAPEOX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2028-10-24 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (mPR) rate | Up to approximately 18 weeks
  mPR rate is defined as the proportion of participants with ≤10% residual viable tumor (RVT) value in the surgical resection sample as determined by local assessment.
Number of participants with adverse events (AEs), serious adverse events (SAEs), immune-mediated adverse events (imAEs), and AEs leading to death or discontinuation of study intervention | Up to approximately 105 weeks

SECONDARY OUTCOMES:
Percentage of participants for whom primary tumour resection is not excluded | Up to approximately 18 weeks
Complete pathologic response (cPR) rate | Up to approximately 18 weeks
  cPR rate is defined as the proportion of participants with 0% RVT value in the surgical resection sample as determined by local assessment.
Major pathological response excluding cPR rate | Up to approximately 18 weeks
  mPR rate is defined as the proportion of participants with ≤10% RVT value in the surgical resection sample as determined by local assessment. cPR rate is defined as the proportion of participants with 0% RVT value in the surgical resection sample as determined by local assessment.
Partial pathologic response rate | Up to approximately 18 weeks
  Partial pathologic response rate is defined as the proportion of participants with >10% and ≤50% RVT value in the surgical resection sample as determined by local assessment.
Negligible pathologic response rate | Up to approximately 18 weeks
  Negligible pathologic response rate is defined as the proportion of participants with >50% RVT value in the surgical resection sample as determined by local assessment.

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (8):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Ostend
  - GSK Investigational Site, Roeselare
- GSK Investigational Site, Udine, Italy
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Geneva, Switzerland
- United Kingdom (3):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Leeds West Yorkshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/